CLINICAL TRIAL: NCT05680246
Title: Prospective Observational Study to Investigate Long-term Outcomes After Prolonged Dual Hypothermic Oxygenated Machine Perfusion of Human Donor Livers (DHOPEPROLONG)
Brief Title: Long-term Outcomes After Prolonged Dual Hypothermic Oxygenated Machine Perfusion of Donor Livers (DHOPEPROLONG)
Acronym: DHOPEPROLONG
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: UMCG_DHOPE-PRO-LONG_2023/01
Record Dates: First submitted 2022-12-25; First posted 2023-01-11 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Liver Transplantation
Keywords: machine preservation; machine perfusion; donor organ preservation; hypothermic oxygenated machine perfusion; donor liver machine perfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DHOPE-PRO: Outcomes of recipients who underwent liver transplantation of donor organs that were perfused with prolonged (>4 hours) DHOPE.
  Interventions: Device: DHOPE-PRO

INTERVENTIONS:
Device: DHOPE-PRO — Prolonged DHOPE preservation >4 hours

SUMMARY:
End-ischemic dual hypothermic oxygenated machine perfusion (DHOPE) of human donor livers mitigates ischemia-reperfusion injury, resulting in a reduction of post-reperfusion syndrome, early allograft dysfunction and biliary complications, when compared with static cold storage. End-ischemic DHOPE can be used to prolong donor liver preservation time for up to 24 hours. According to IDEAL-D (Idea, Development, Exploration, Assessment, Long term study-Framework for Devices), scientific evidence for prolonged DHOPE has currently reached stage 3. Assessment of long-term outcomes after prolonged DHOPE preservation based on real-world data (i.e., IDEAL-D stage 4) is currently still lacking.

DETAILED DESCRIPTION:
The aim of this study is to assess long-term outcomes after transplantation of donor livers preserved by prolonged hypothermic oxygenated machine perfusion (DHOPE-PRO).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years) who underwent liver transplantation of donor livers preserved with end-ischemic DHOPE for >4 hours

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult liver transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Death-censored graft survival | Up to 5-years
  Death-censored graft survival, assessed by survival analysis methods.

SECONDARY OUTCOMES:
Overall graft survival | Up to 5-years
  Overall graft survival, assessed by survival analysis methods.
overall patient survival | Up to 5-years
  overall patient survival, assessed by survival analysis methods.
arterial and biliary complication-free survival (ABCFS) | Up to 5-years
  arterial and biliary complication-free survival (ABCFS), assessed by survival analysis methods.
incidence of biliary complications | Up to 5-years
  incidence of biliary complications
incidence of vascular complications | Up to 5-years
  incidence of vascular complications
incidence of acute cellular rejection | Up to 5-years
  incidence of acute cellular rejection
incidence of chronic rejection | Up to 5-years
  incidence of chronic rejection
incidence of re-transplantation | Up to 5-years
  incidence of re-transplantation
incidence of recurrence of primary disease | Up to 5-years
  incidence of recurrence of primary disease (including recurrence of malignancies)
incidence of new-onset chronic kidney disease | Up to 5-years
  incidence of new-onset chronic kidney disease
incidence of new-onset diabetes after transplantation | Up to 5-years
  incidence of new-onset diabetes after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Vincent E de Meijer, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared upon reasonable request, only with appreciation of the national and local institute's privacy regulations